CLINICAL TRIAL: NCT05292846
Title: Uninterrupted Direct-acting Oral Anticoagulation in Patients Undergoing Transradial Percutaneous Coronary Procedures
Acronym: DOAC-NOSTOP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Jorge Sanz Sanchez, Principal Investigator, Hospital Universitario La Fe
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 515
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease; Bleeding; Direct Acting Anticoagulant Adverse Reaction
MeSH Terms: conditions — Coronary Artery Disease; Hemorrhage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Uninterruped direct-acting oral anticoagulation (Experimental): Uninterrupted direct-acting oral anticoagulation in patients undergoing trans-radial percutaneous coronary procedures
  Interventions: Drug: Direct-acting oral anticoagulation

INTERVENTIONS:
Drug: Direct-acting oral anticoagulation — Apixaban Dabigatran Edoxaban Rivaroxaban

SUMMARY:
Up to 20-30% of patients who are candidates for direct oral anticoagulation (DOAC) present with concomitant ischemic heart disease and often require coronary angiography with or without percutaneous coronary intervention (PCI). The decision whether to continue the DOAC throughout periprocedural period or interrupt DOAC before planned procedure represents a substantial challenge in daily clinical practice.

The objective of this study is to evaluate the safety of uninterrupted direct-acting oral anticoagulation in patients undergoing trans-radial percutaneous coronary procedures.

DETAILED DESCRIPTION:
The study design is an investigator-initiated, single-arm, open-label, pilot study in patients treated with DOAC undergoing trans-radial percutaneous coronary procedures.

Because of the exploratory nature of this study, no formal sample size calculations are required. On the basis of previous pilot studies with similar designs, a sample of 200 patients is planned; with a safety stopping rule based on the occurrence of BARC type 3 or 5 bleeding. In the present trial, if during the enrollment period more than 3 cases of BARC 3 or 5 bleeding occur up to 30-day follow-up, patient recruitment will be terminated. This number is based on the reported 1.6% BARC type 3 or 5 bleeding in patients undergoing transradial percutaneous coronary procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients under anticoagulation with DOAC and any indication for diagnostic or therapeutic trans-radial percutaneous coronary procedures. At least 25% of the population undergoing PCI will be included.

Exclusion Criteria:

1. Aged < 18 years
2. Cardiogenic shock
3. Major active bleeding at the time of the procedure
4. Use of mechanical circulatory support
5. Chronic total occlusions
6. Pre-planned vascular access different from radial artery access (i.e. femoral, brachial, ulnar)
7. Inability to provide informed consent
8. Unable to understand and follow study-related instructions or unable to comply with study protocol
9. Currently participating in another trial
10. Pregnant women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
Rate of Bleeding Academic Research Consortium (BARC) type 2, 3 or 5 | 30-day follow-up

SECONDARY OUTCOMES:
Rate of BARC type 3, or 5 | 30-day follow-up
Rate of all-cause death | 30-day follow-up
Rate of cardiac death | 30-day follow-up
Rate of stroke | 30-day follow-up
Rate of myocardial infarction | 30-day follow-up
Rate of definite/probable stent thrombosis | 30-day follow-up
Rate of definite stent thrombosis | 30-day follow-up
Rate of target-lesion revascularization | 30-day follow-up
Rate of target-vessel revascularization | 30-day follow-up

CONTACTS AND LOCATIONS:
Locations (4):
- Humanitas Research Hospital, Rozzano, Milan, Italy
- Spain (3):
  - Hospital del Mar, Barcelona
  - Hospital La Paz, Madrid
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study will be available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Valgimigli M, Frigoli E, Leonardi S, Rothenbuhler M, Gagnor A, Calabro P, Garducci S, Rubartelli P, Briguori C, Ando G, Repetto A, Limbruno U, Garbo R, Sganzerla P, Russo F, Lupi A, Cortese B, Ausiello A, Ierna S, Esposito G, Presbitero P, Santarelli A, Sardella G, Varbella F, Tresoldi S, de Cesare N, Rigattieri S, Zingarelli A, Tosi P, van 't Hof A, Boccuzzi G, Omerovic E, Sabate M, Heg D, Juni P, Vranckx P; MATRIX Investigators. Bivalirudin or Unfractionated Heparin in Acute Coronary Syndromes. N Engl J Med. 2015 Sep 10;373(11):997-1009. doi: 10.1056/NEJMoa1507854. Epub 2015 Sep 1. PMID 26324049
- [Result] Lip GY, Huber K, Andreotti F, Arnesen H, Airaksinen KJ, Cuisset T, Kirchhof P, Marin F; European Society of Cardiology Working Group on Thrombosis. Management of antithrombotic therapy in atrial fibrillation patients presenting with acute coronary syndrome and/or undergoing percutaneous coronary intervention/ stenting. Thromb Haemost. 2010 Jan;103(1):13-28. doi: 10.1160/TH09-08-0580. Epub 2009 Sep 30. PMID 20062939
- [Result] Kogame N, Guimaraes PO, Modolo R, De Martino F, Tinoco J, Ribeiro EE, Kawashima H, Ono M, Hara H, Wang R, Cavalcante R, Moulin B, Falcao BAA, Leite RS, de Almeida Sampaio FB, Morais GR, Meireles GC, Campos CM, Onuma Y, Serruys PW, Lemos PA. Aspirin-Free Prasugrel Monotherapy Following Coronary Artery Stenting in Patients With Stable CAD: The ASET Pilot Study. JACC Cardiovasc Interv. 2020 Oct 12;13(19):2251-2262. doi: 10.1016/j.jcin.2020.06.023. Epub 2020 Sep 16. PMID 32950419
- [Result] Serruys PW, van Hout B, Bonnier H, Legrand V, Garcia E, Macaya C, Sousa E, van der Giessen W, Colombo A, Seabra-Gomes R, Kiemeneij F, Ruygrok P, Ormiston J, Emanuelsson H, Fajadet J, Haude M, Klugmann S, Morel MA. Randomised comparison of implantation of heparin-coated stents with balloon angioplasty in selected patients with coronary artery disease (Benestent II). Lancet. 1998 Aug 29;352(9129):673-81. doi: 10.1016/s0140-6736(97)11128-x. PMID 9728982
- [Result] Lip GYH, Collet JP, Haude M, Byrne R, Chung EH, Fauchier L, Halvorsen S, Lau D, Lopez-Cabanillas N, Lettino M, Marin F, Obel I, Rubboli A, Storey RF, Valgimigli M, Huber K; ESC Scientific Document Group. 2018 Joint European consensus document on the management of antithrombotic therapy in atrial fibrillation patients presenting with acute coronary syndrome and/or undergoing percutaneous cardiovascular interventions: a joint consensus document of the European Heart Rhythm Association (EHRA), European Society of Cardiology Working Group on Thrombosis, European Association of Percutaneous Cardiovascular Interventions (EAPCI), and European Association of Acute Cardiac Care (ACCA) endorsed by the Heart Rhythm Society (HRS), Asia-Pacific Heart Rhythm Society (APHRS), Latin America Heart Rhythm Society (LAHRS), and Cardiac Arrhythmia Society of Southern Africa (CASSA). Europace. 2019 Feb 1;21(2):192-193. doi: 10.1093/europace/euy174. PMID 30052888
- [Derived] Sanz-Sanchez J, Chiarito M, Calderon AT, Santos IA, Cao D, Jurado-Roman A, Montilla BV, Tartaglia F, Garrido PP, Nardin M, Romero JS, Vallinas-Hernandez S, Marquez DT, Carrasco-Moraleja M, Reimers B, Dolz LM, Diez-Gil JL, Stefanini G, Garcia-Garcia HM. Uninterrupted Direct-Acting Oral Anticoagulation in Patients Undergoing Transradial Percutaneous Coronary Procedures: The DOAC-NOSTOP. Catheter Cardiovasc Interv. 2025 Aug;106(2):1371-1377. doi: 10.1002/ccd.31691. Epub 2025 Jun 18. PMID 40530906